CLINICAL TRIAL: NCT07215195
Title: Neuropsychiatric Outcomes and Disrupted Sleep Following Acquired Brain Injury
Acronym: NODS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID 18842
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-07

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: stroke; traumatic brain injury; neuropsychiatric disorder; movement; sleep; brain injury
MeSH Terms: conditions — Brain Injuries; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with acquired brain injury: We will follow adults with either stroke or traumatic brain injury for one year post-injury to examine the associations between sleep, mental health and motor recovery.

SUMMARY:
The two most common causes of brain injury are stroke and trauma. Both sleep and mental health problems are common after brain injury; we will investigate whether there is a relationship between poor sleep quality and worse mental health in this group. We will also follow patients up, at approximately three-monthly intervals until one year after injury, to see how sleep and mental health symptoms change over time and with recovery.

We will assess sleep in detail using questionnaires, a sleep monitor worn on the wrist, a portable brain activity sensor, and a sleep mat. We will assess mental health (neuropsychiatric) symptoms using questionnaires.

Participants will be asked to complete these assessments at baseline and at approximately 3-monthly intervals until they reach 12 months post-injury.

This data will allow us to explore the types of sleep disruption seen after brain injury and examine the association between sleep and mental health symptoms.

DETAILED DESCRIPTION:
This is a cross-sectional and longitudinal observational cohort study to assess the relationship between sleep quality and neuropsychiatric symptoms in adults within 12 months of an acquired brain injury, including traumatic brain injury (TBI), ischaemic stroke or haemorrhage. We hypothesise that participants with poor sleep quality will have worse neuropsychiatric (mental health) symptoms and slower recovery.

Participants will be identified at least one week, but less than 12 months, after brain injury from: a) National Health Service (NHS) sites; b) advertisements; and c) previous studies where patients have consented to be contacted about future studies.

The primary aim is to test whether adults with acquired brain injury and poor sleep quality (defined as a cut-off of >5 on the Pittsburgh Sleep Quality Index; PSQI) have a greater neuropsychiatric symptom burden (assessed with the diagnostic and statistical manual of mental disorder ver sion (DSM-5) Cross-Cutting Measure Level 1 Total Score) than those with good subjective sleep quality.

Secondary outcomes will test whether both self-reported and objective markers of sleep disruption (derived from actigraphy, brain activity and sleep mat data) relate to neuropsychiatric symptoms over time.

Two optional sub-studies will assess: a) long term sleep mat derived metrics (the participant will be asked to have a sleep mat on their bed at home for one year), and b) the association between sleep and changes in motor function over time.

Baseline clinical and demographic characteristics will be gathered from medical records and/or using questionnaires.

For the main objective of the study (cross-sectional assessment), we will collect data at a single time point (baseline). Following informed consent, we will assess sleep quality using the Pittsburgh Sleep Quality Index questionnaire (PSQI) and Neuropsychiatric symptoms using the Diagnostic and Statistical Manual (DSM-5) Cross-Cutting measure (DSM-5 CCM) level 1 total score.

For the secondary objectives, we will collect data at as many time points as the participant is able and willing to complete. Assessments will be at 3-monthly intervals until the participant reaches 12 months post-injury, thus some participants will complete more assessments than others. Secondary measures regarding sleep and neuropsychiatric symptoms will be assessed with self-report questionnaires at each time point: Pittsburgh Sleep Quality Index questionnaire (PSQI), sleep diary (SD; daily for 2 weeks), insomnia severity index (ISI), Fatigue Severity Scale (FSS), patient health questionnaire (PHQ-8), generalized anxiety disorder questionnaire (GAD-7), DSM-5 Cross-Cutting measure (DSM-5 CCM) Level 1 (total), primary care post-traumatic stress disorder questionnaire (PC-PTSD). We will also obtain information regarding the patient's location at the time of assessment (e.g. hospital, neurorehabilitation unit, home), medications and any sleep or mental health treatments they have received.

We will collect 'objective' sleep measures which will include using a waterproof actigraphy monitor worn on the least-affected wrist (2 weeks at each assessment period), a portable brain activity (electroencephalography) monitor to wear on their head during sleep (3-5 nights at each timepoint) and a sleep mat which goes under the bed mattress (2 weeks at each timepoint).

There are two optional sub-studies:

1. For a subset of participants we will provide a sleep mat to keep under their mattress continuously until they reach 12 months post-injury. This is to explore changes in sleep continuity/disruption and sleep timing long-term.
2. For a subset of participants we will assess motor impairment/function of the upper limb (arm) and lower limb (leg) at each time point using clinical/research assessments: the Fugl Meyer assessment, Action Research Arm Test, Box and Blocks test, and the Rivermead Mobility Index.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* At least one week, but less than 12 months post-injury
* Clinical diagnosis of acquired brain injury (stroke, haemorrhage or traumatic).
* Participants with Traumatic Brain Injury will have a Mild (probable) or Moderate-severe (definite) brain injury according to the Mayo classification
* Participants must be willing to consent to us contacting their general practitioner (GP) or direct care team if we have concerns about their mental health

Exclusion Criteria:

* Brain injury not caused by trauma, haemorrhage or stroke
* Previous brain injury.
* Other relevant neurological conditions which could affect outcome measures (e.g., Parkinson's or Alzheimer's disease)
* No stable and suitable place to sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, age 18 years or over (no upper age limit) within one year of acquired brain injury (stroke, haemorrhage, trauma)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric (mental health) symptoms at baseline | Baseline (first assessment, obtained within 12 months of acquired brain injury)
  Assessed using the Diagnostic and Statistical Manual version 5 (DSM-5) Cross-Cutting Measure questionnaire level 1 total score. Range 0-92, higher scores indicate worse neuropsychiatric symptoms.
Self reported sleep quality at baseline | Baseline (first assessment, obtained within 12 months of acquired brain injury)
  Assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Range 0-21, higher scores indicate worse sleep quality.

SECONDARY OUTCOMES:
Neuropsychiatric (mental health) symptoms | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Diagnostic and Statistical Manual version 5 (DSM-5) Cross-Cutting Measure questionnaire level 1 total score. Range 0-92, higher scores indicate worse neuropsychiatric symptoms.
Sleep Fragmentation Index | Baseline, and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using actigraphy (wearable activity monitor) over two weeks. Higher values indicate more disrupted (worse) sleep. The minimum value is 0. There is no specified maximum value. According to the manual for the software which does the calculation the definition of sleep fragmentation index is "the sum of the Mobile time (%)' and the 'Immobile bouts <=1min".There are no units associated with sleep fragmentation.
Time in each stage of sleep | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Electroencephalography (EEG) headband for assessing sleep measures over 3 nights. Time spent in each stage of sleep, in minutes as a percentage of the total sleep time. Stages include Non-rapid eye movement (NREM) sleep 1, 2 and 3. Range 0-100%
Slow wave sleep (SWS) amplitude | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed with electroencephalography over 3 nights. Amplitude, in microvolts. Minimum value 0, there is no specified maximum value. Higher values indicate larger (higher amplitude) slow wave oscillations in the brain.
Sleep spindle power | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed with electroencephalography over 3 nights. Power, in decibels. Minimum value 0, no specified maximum value. Higher values indicate higher power of the sleep spindle frequency brain activity.
Sleep continuity measures from a mattress sensor | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Sleep measures assessed using Withing's sleep analyser under-mattress sensor over a two week period (e.g. apnea episodes, time in each sleep stage, sleep duration, sleep fragmentation).
Symptoms of Depression | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using the Patient Health Questionnaire (8-item), range 0-24 (higher values indicate more depressive symptoms)
Symptoms of Anxiety | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using the Generalised Anxiety Disorder - 7 item (GAD-7) questionnaire. Scores range from 0-21, higher values indicate more anxiety symptoms.
Symptoms of Post-traumatic stress disorder | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed with the Primary Care Screen for DSM-5 (PC-PTSD-5), scores range from 0-5, higher values indicate more severe postraumatic stress disorder symptoms.
Symptoms of Insomnia | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using the Insomnia Severity Index (ISI) questionnaire. Range 0-28, higher scores indicate more severe symptoms of insomnia.
Self reported sleep quality | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Range 0-21, higher scores indicate worse sleep quality.
Fatigue symptoms | Baseline and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using the Fatigue Severity Scale (FSS) questionnaire. Scores range from 0-63, higher values indicate worse fatigue.
Sleep Regularity Index | Baseline, and at 3-monthly intervals until the patient reaches 12 months following acquired brain injury (up to 4 assessments per participant).
  Assessed using actigraphy (wearable activity monitor) over two weeks. Score 0-100, higher values indicate more regular sleep-wake patterns. There are no units associated with the sleep regularity index.

OTHER OUTCOMES:
Sleep continuity assessed with a mattress sensor | Continuous from baseline until 12 months after acquired brain injury
  Time-series (longitudinal) assessment of sleep measures using the Withings under mattress sleep sensor kept in place for the duration of the study (e.g. (e.g. apnea episodes, time in each sleep stage, sleep duration, sleep fragmentation).
Motor impairment | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Fugl Meyer Assessment. Range 0-100, lower score indicates worse motor impairment
Upper limb ability | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Action Research Arm Test. Range 0-57, higher score indicates better upper limb ability
Hand function | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Box and Blocks Test, as the number of blocks moved in 60 seconds. Minimum value 0, no specified maximum value. Higher score indicates better hand function.
Mobility | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Rivermead Mobility Index. Range 0-15, higher score indicates better functional mobility
Estimated total sleep time | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using actigraphy (wearable activity monitor) over a two-week period. Time, in minutes. Higher values indicate longer sleep time
Wake After Sleep Onset (WASO) | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using actigraphy (wrist worn activity monitor) over two weeks. Time, in minutes. Minimum value=0, no maximum value. Higher value indicates worse sleep
Sleep efficiency | Baseline, and at 3-monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using actigraphy (wrist worn activity monitor) over two-weeks. Score is the percentage of time in bed spent asleep. Range 0-100%. Lower sleep efficiency indicates worse sleep
Subjective sleep diary measures | Baseline, and at 3 monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using sleep diary data collected over two weeks (e.g. estimated time to get into bed, sleep onset latency, total sleep time, wake after sleep onset, rise time).
Current and past psychiatric disorder at baseline | Baseline (first assessment, within 12-months of acquired brain injury)
  Assessed using a brief questionnaire based on ICD-11 criteria for depression, generalised anxiety disorder, panic disorder, obsessive compulsive disorder, agoraphobia, adjustment disorder, bipolar disorder and psychosis.
Presence of Sleep Disorders | Baseline, and at 3 monthly intervals until 12 months following injury (up to 4 assessments per participant)
  Assessed using the Sleep Disorders Screening questionnaire. Positive responses within sub-groups of questions indicate potential presence of specific sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fleming, PhD, Principal Investigator — University of Oxford
Locations (1):
- Wellcome Centre for Integrative Neuroimaging (WIN) FMRIB, Nuffield Department of Clinical Neurosciences, John Radcliffe Hospital, Oxford OX3 9DU, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be available upon reasonable request to Melanie Fleming
Time Frame: Data will be available following publication or public release of the main findings, for approximately 2 years.
Access Criteria: Anonymous data will be available upon reasonable request to the Principal Investigator, using file transfer (e.g. Microsoft OneDrive).